CLINICAL TRIAL: NCT04390191
Title: Early Continuous Positive Airway Pressure (CPAP) in COVID-19 Confirmed or Suspected Patients
Brief Title: Early CPAP in COVID-19 Confirmed or Suspected Patients
Acronym: PAP-COVID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Declining cases of COVID in New York due to vaccinations and new treatments for outpatient management
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Itamar-Medical, Israel (Industry); Community Surgical Supply of Toms River, Inc (Industry); Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Neomi A Shah, Associate Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-0900
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; COVID; Coronavirus
Keywords: Continuous Positive Airway Pressure; COVID-19; Coronavirus; Positive airway pressure; Hospital admission; Non-invasive ventilation
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, parallel group, open-label, randomized clinical trial, where the study team will investigate the efficacy of continuous positive airway pressure therapy (CPAP) in COVID suspected or confirmed patients who are sent home from the emergency room with mild pneumonia or respiratory illness but who do not require hospital admission. The study team proposes a randomized controlled trial of CPAP (n=100) vs. control (n=100) in COVID-19 suspected or confirmed patients with pneumonia or respiratory illness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Continuous Positive Airway Pressure (CPAP) (Experimental): Patients will be given CPAP at fixed pressure of 8-10 cm water pressure for 72 hours continuously
  Interventions: Device: Continuous Positive Airway Pressure
- Control (No Intervention): Patients in this arm will be not be given any intervention and will be monitored for 72 hours continuously, and then daily for a total of 14 days.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — CPAP at fixed pressure (8-10cm H20) for 72 hours continuously (except for daily activities such as eating, personal activities and breaks for ambulation etc).
  Other Names: CPAP
  Arms: Continuous Positive Airway Pressure (CPAP)

SUMMARY:
There is surge in COVID infected patients in New York City with a shortage of hospital beds, ICU beds and ventilators. Strategies to reduce the need for all of the above are immediately needed. Further, few interventions are targeted in COVID infected patients early in the course of their disease and especially in the community/home settings. Respiratory decompensation appears to occur later in the disease process (i.e. 7-10 days after becoming symptomatic) therefore many patients are sent home from the Emergency Room and they subsequently decompensate later at home. Some patients die at home and others are returning to the Emergency Room with hypoxemic respiratory failure. There is no treatment offered to this population of patients, i.e. COVID suspected or confirmed and with respiratory symptoms or abnormal chest x-ray at the time of presentation. Based on experience across the globe, these patients are likely to worsen at home. The study team therefore proposes a prospective, single-center, parallel group, open-label, randomized clinical trial to assess the efficacy of fixed low continuous positive airway pressure therapy (CPAP) (FDA approved and often used for treatment of sleep apnea) in COVID confirmed or suspected patients with abnormal chest x-ray or respiratory symptoms who do not require hospital admission and are discharged home from the emergency room.

DETAILED DESCRIPTION:
The study team proposes a randomized controlled trial of CPAP (n=100) vs. control (n=100) in COVID-19 suspected or confirmed patients with pneumonia or respiratory illness. The overarching aim of this proposal is to determine if early use of CPAP at home will reduce hypoxemic events or reduce the need for hospital admission or death in COVID-19 suspected or confirmed patients. The study team will include adult patients (age>18) who live alone or have more than one bedroom at home, with serologically confirmed or suspected COVID-19 infection, who have one or more of the following: fever (>38ºC), sore throat, myalgia or flu-like illness AND have one or more of the following additional symptom or diagnostic criteria: abnormal chest x-ray, new onset cough, mild hypoxemia at rest (saturation less than 96%), abnormal lung exam, chest tightness or shortness of breath AND who are without need for hospital admission. Patients with preexisting pulmonary diseases such as advanced COPD, advanced parenchymal lung disease, history of pneumothorax etc. will be excluded. Participants in both arms will be shipped a pulse oximeter to monitor oxygen saturation and a disposable home sleep apnea monitor (WatchPAT) to track blood oxygen level continuously for 12 hours with data feed into a cloud based platform. Additionally, 100 patients will be randomized to receive CPAP at fixed pressure (8-10cm H20) for 72 hours continuously (except for daily activities such as eating, personal activities and breaks for ambulation etc). The CPAP pressure will be adjusted based on patient's comfort but will not deviate from the range of 8-10cm. While the study protocol will end at 72 hours, patients who wish to continue CPAP will be allowed to do so for symptomatic benefit up to 7 days from randomization. All CPAP recipients will be given a full-face mask and will be asked to stay in quarantine for the duration of the protocol to avoid risk of infecting family members with aerosol (separate consent to be obtained from household members who are elderly or with comorbidities.) The study team hypothesizes that early low-grade fixed CPAP in COVID infected patients who have respiratory abnormalities will reduce hypoxemic events and decrease the risk of subsequent hospitalization or death in 14 days from randomization. The study will also address whether use of CPAP in the home increases the risk of infecting household family members.

ELIGIBILITY:
Inclusion criteria:

1. Adults > 18 years old
2. Patients living alone or with more than one room at home
3. COVID confirmed or suspected
4. To be discharged home or already discharged
5. One or more of these: fever (>38oC), sore throat, myalgia or flu-like illness
6. One or more of the following: abnormal chest x-ray, new onset cough, mild hypoxemia (saturation between 92-96%), abnormal lung exam, chest tightness or shortness of breath

Exclusion criteria:

1. Unable to self quarantine for 72 hours if in the CPAP arm
2. Preexisting pulmonary diseases such as advanced COPD, advanced parenchymal lung disease, history of pneumothorax etc.
3. Claustrophobic and unable to tolerate CPAP mask
4. Evidence of hypercapnia
5. Recent heart of lung surgery within 3 months
6. Individuals without access to smart phones or wireless connection or internet access
7. Prior history of aspiration
8. Speech or swallowing impairment (risk of aspiration)
9. History of stroke with significant neurologic deficit
10. Advanced symptomatic heart failure
11. Unable to provide informed consent
12. household with young children and child care responsibilities
13. household with high-risk individuals (defined as over 60 or with comorbidities (e.g. heart disease, diabetes, pulmonary))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neomi Shah, MD, MPH, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period from May 2020 to July 2021
Groups:
- Control: Patients in this arm was not be given any intervention and will be monitored for 72 hours continuously, and then daily for a total of 14 days.
Period: Overall Study
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Started | 1 | 3
Completed | 0 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (0) | 54.67 (12.01) | 48.50 (15.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Met the Efficacy Endpoint
Description: Number of participants who met the efficacy endpoint within 14 days. The efficacy endpoint is meeting any of the following: All-cause mortality within 14 days of randomization, hospital admission (including ED visit) within 14 days of randomization, oxygen saturation less than 90 during the 72-hour observation period from randomization, absolute reduction in oxygen saturation of more than 4% during the 72-hour observation period from randomization.
  If a participant meets any of the events noted in the composite endpoint, it is counted as a worse outcome. The composite endpoints were selected based on available covid-related information at the time of the study design. This study was conducted to determine measures that alleviated hospital burden, allowing patients to be managed at home. Oxygen-related endpoints measure improvement in a home setting and contribute to a higher number of events in the composite outcomes, to provide enough power to measure efficacy in a small trial.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 1 | 3
Participants | 1 | 0

2. Secondary Outcome: Number of Participants Admitted to the ICU
Description: Number of Participant with an admission to the intensive care unit within 14 days from randomization
Time Frame: 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 1 | 3
Participants | 0 | 0

3. Secondary Outcome: Time to Intubation and Mechanical Ventilation
Description: The time from randomization to the patient needing to be intubated and needing mechanical ventilation within 14 days from randomization
Time Frame: 14 days from randomization
Population: No participants intubated.
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Deaths at 14 Day and 28 Day Mortality
Description: Mortality Rate - the number of deaths within 14 and 28 days from randomization
Time Frame: 14-28 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 1 | 3
Participants
  14 days after randomization | 0 | 0
  28 days after randomization | 0 | 0

5. Secondary Outcome: Conversion of COVID Household Members in CPAP vs Control
Description: The number of household members converting from being COVID negative to COVID positive in the CPAP arm vs the control arm within 14 days from randomization
Time Frame: 14 days from randomization
Measure: Number; unit: household members
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 1 | 3
household members | 0 | 0

6. Secondary Outcome: Change in Clinical COPD Questionnaire (CCQ)
Description: Mean Change in CCQ - If there is any improvement in respiratory symptoms of cough or shortness of breath etc. assessed via a respiratory symptom questionnaire within 14 days from randomization. Patients were monitored for 72 hours continuously, and then daily for a total of 14 days. The time frame is a change between the baseline COPD score at the time of enrollment and the last COPD score recorded within the following 14 days.
  The CCQ is a 10-item instrument questionnaire, with each question scored on a scale of 0 to 6. Thus, the full scale is 0 to 60, with higher score indicating lower health status. A negative value indicates that their score improved. A decrease in CCQ indicates improvement, Last Observation Carried Forward (LOCF) applied.
Time Frame: baseline and 14 days from randomization
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 1 | 3
score on a scale | -11 | 4.6 [-5 to 15]

7. Secondary Outcome: Number of Patients Electing to Continue CPAP for Greater Than 72 Hours
Description: Number of the patients in the CPAP arm elect to continue using the CPAP after the initial 72 hour period.
Time Frame: 7 days from randomization
Population: CPAP arm only
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 1 | 0
Participants | 1 |

8. Secondary Outcome: Number of Participants With Improvement in Oxygen Saturation
Description: The number of participants with improvement in oxygen saturation within 14 days of randomization.
Time Frame: 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 1 | 3
Participants | 0 | 1

9. Secondary Outcome: Number of Participants With Hospital Admission or ED
Description: Number of participants with hospital admission or ED within 14 days of randomization
Time Frame: 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
Number analyzed (Participants) | 1 | 3
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 28 days. Patients were followed for 28 days and as a secondary endpoint, we assessed 28 day mortality and for late impact of CPAP.
Description: The control subject who was admitted to the ER for an adverse event still completed the study. The subject was routinely contacted and completed study questionnaires. The adverse event was considered as an outcome and he was not withdrawn from the study.
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Positive Airway Pressure (CPAP) (N=1) | Control (N=3)
COVID pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Subject was admitted to ER for worsening symptoms of COVID-19, including Covid pneumonitis with SOB, fever, and diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT04390191/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT04390191/SAP_001.pdf